CLINICAL TRIAL: NCT03557008
Title: Systems Biology of Inactivated Rabies Vaccine in Healthy Adults With or Without Use of Broad Spectrum Antibiotics
Brief Title: Responses to Rabies Vaccine in Adults With or Without Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00101567
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Rabies Human
Keywords: Rabies Vaccine; Antibiotics; Biopsy
MeSH Terms: interventions — Rabies Vaccines; Metronidazole; Vancomycin; Neomycin

STUDY DESIGN:
Intervention Model Description: Longitudinal and Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rabies Vaccine with Antibiotics (Active Comparator): Participants in this group will receive the rabies vaccines as well as an antibiotic regimen consisting of metronidazole, vancomycin, and neomycin sulfate.
  Interventions: Biological: Rabies Vaccine; Drug: Metronidazole; Drug: Vancomycin; Drug: Neomycin Sulfate
- Rabies Vaccine (Active Comparator): Participants in this group will receive the rabies vaccine.
  Interventions: Biological: Rabies Vaccine

INTERVENTIONS:
Biological: Rabies Vaccine — A 1.0 milliliter (mL) dose of Imovax® will be given to participants on Day 0 and Day 28 of the study.
  Other Names: Imovax
Drug: Metronidazole — The antibiotic regimen will be given for five days beginning 3 days prior to vaccination, on the vaccination day, and one day after vaccination for a total for 5. The regimen will include 500 milligrams (mg) of Flagyl taken by mouth three times a day.
  Other Names: Flagyl
  Arms: Rabies Vaccine with Antibiotics
Drug: Vancomycin — The antibiotic regimen will be given for five days beginning 3 days prior to vaccination, on the vaccination day, and one day after vaccination for a total for 5. The regimen will include 125 mg of Vancocin taken by mouth four times a day.
  Other Names: Vancocin
  Arms: Rabies Vaccine with Antibiotics
Drug: Neomycin Sulfate — The antibiotic regimen will be given for five days beginning 3 days prior to vaccination, on the vaccination day, and one day after vaccination for a total for 5. The regimen will include 500 milligrams (mg) of Neomycin sulfate taken by mouth three times a day.
  Other Names: Mycifradin
  Arms: Rabies Vaccine with Antibiotics

SUMMARY:
The use of antibiotics changes micro-organisms in the intestines which may impact the body's vaccine immune response and alter the effectiveness of the rabies vaccine.

There will be two randomized groups (1:1 randomization). Group A will start taking an antibiotic regimen by mouth 3 days prior to vaccination and continue taking antibiotics the day of rabies vaccination and one day after vaccination for a total of 5 days. Group B will only receive the rabies vaccination and will not take any antibiotics. The dosage of each antibiotic is taken from their respective package inserts and does not exceed the maximum dose allowed for each antibiotic.

The purpose of the study is to look at immune response after rabies vaccination with or without the use of antibiotics from day of vaccination to 28 days post vaccination in both groups.

DETAILED DESCRIPTION:
Vaccination has been one of the most important and cost-effective public health interventions to provide protection against infectious diseases. Since the introduction of the first vaccine in 1796, there have been countless advances in the field. However, numerous gaps remain to be addressed. An important gap is understanding the mechanisms that lead to suboptimal immune responses to vaccination. It has been shown that the magnitude of the immune response produced by vaccines is highly variable among individuals, with both genetic and environmental factors playing an important role. More recently, emphasis is being placed on the role of the microbiota in vaccine immunogenicity. The microbiome is the collection of all microbial cells in and on the human body, with the majority being in the gastrointestinal tract. The composition of the microbiome has the ability to affect B and T cell development, which are important aspects of the adaptive immune system and major responders to vaccination.

Due to this link between microbiome and the immune system, it is important to further understand the impact of the microbiome on the immune response to vaccination. This can be done using systems vaccinology, which is the application of systems biology in vaccinology to predict vaccine efficacy. The aim is to find molecular signatures, or patterns of gene expression induced after vaccination, which can be used to correlate and predict the development of protective immunity. The goal of this study is to determine whether alteration of microbiota by antibiotic exposure can negatively impact the immunogenicity of rabies vaccine, and to assess the innate and adaptive immune mechanisms responsible for that phenomenon.

Half of the study participants will receive the rabies vaccine alone and half will receive the rabies vaccine along with a 5 day course of antibiotics. The primary objective of this study is to compare antibody titers 28 days after vaccination with the rabies vaccine in adults with or without use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-49 years.
* Able to understand and give informed consent.
* Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for 28 days before and 28 days after Rabies vaccination.

Exclusion Criteria:

* Receipt of the following:

  * Receipt of blood products 3 months prior to vaccination or expected receipt through 12 months after vaccination.
  * Receipt of any live virus vaccines within 28 days prior to vaccination or expected receipt within 28 days after vaccination.
  * Receipt of any inactivated vaccine within 14 days or expected receipt within 14 days after vaccination.
  * Receipt of any antibiotic 3 months prior to vaccination or expected receipt 28 days after vaccination.
  * Receipt of probiotics and prebiotics 3 months prior to vaccination or expected receipt 28 days after vaccination.
  * Receipt of proton pump inhibitors, H2 receptor blockers, or antacids 3 months prior to vaccination or expected receipt 28 days after vaccination.
* Presence of co-morbidities or immunosuppressive states such as:

  * Chronic medical problems including (but not limited to) insulin dependent diabetes, severe heart disease (including arrhythmias), severe lung disease, auto immune diseases, thrombocytopenia and grade 4 hypertension. Grade 4 hypertension per CTCAE criteria is defined as Life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive).
  * Chronic neurologic conditions including seizure disorder, Parkinson's disease, myasthenia gravis, neuropathy, or history of encephalopathy, meningitis or ototoxicity.
  * Any history of gastrointestinal disease including (but not only): documented bacterial gastroenteritis or gastroenteritis associated with fever or associated with presence of blood/mucus in stools in the last 3 months, inflammatory bowel disease, and/or gastrointestinal surgery.
  * Any history of kidney or liver diseases.
  * Alcohol abuse, drug abuse, or psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
  * Any history of lymphoma involving axillary nodes or any history of breast cancer.
  * Impaired immune function or known chronic infections including, but not limited to, known HIV, tuberculosis, hepatitis B or C; organ transplantation (bone marrow, hematopoietic stem cell, or solid organ transplant); immunosuppression due to cancer; current and/or expected receipt of chemotherapy, radiation therapy, steroids (i.e., more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 90 days, or high dose inhaled corticosteroids); and any other immunosuppressive therapies, functional or anatomic asplenia, or congenital immunodeficiency. Subjects receiving > 20 mg/day of prednisone or its equivalent daily or on alternate days for more than 2 weeks may enter the study after therapy has been discontinued for more than 3 months and Subjects are excluded if on high dose intranasal steroids defined as > 960 mcg/day of beclomethasone dipropionate or equivalent.
  * Pregnancy or breast feeding
* Conditions that could affect the safety of the volunteers, such as:

  * Severe reactions to prior vaccinations, including anaphylaxis
  * History of Guillain-Barré syndrome
  * History of bleeding disorders or current use of warfarin, aspirin, heparin, nonsteroidal anti-inflammatory drugs (NSAIDs) or other blood thinner/anticoagulant medications in the past week (for subjects undergoing lymph node sampling)
  * Use of anticonvulsants
  * Use of digoxin or other forms of digitalis
  * Any allergy to any component of the vaccine or lidocaine (for subjects undergoing lymph node sampling)
  * Allergy to vancomycin, metronidazole or neomycin as well as other aminoglycosides (gentamicin, tobramycin, amikacin, streptomycin)
* Volunteers with any acute illness, including any fever within 3 days prior to vaccination.
* Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.
* Positive C difficile testing by polymerase chain reaction (PCR) at screening or history of C difficile infection.
* Any grade 2 safety lab test results at screening
* Previously received any rabies vaccine or immunoglobulin.
* Are at high risk of exposure to rabies: veterinarians, animal handlers, rabies laboratory workers, spelunkers, frequent contact with rabies virus or with possibly rabid animals, international travelers who are likely to come in contact with animals in parts of the world where rabies is common, and rabies biologics production workers.
* Bilateral inflammatory process of upper arms in the past 2 weeks.
* Prior breast or axillary biopsy and/or surgery.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began July 5, 2018 and all follow up for the primary outcome measure was complete by June 2, 2022. Participants were enrolled at the Hope Clinic of the Emory Vaccine Center in Atlanta, Georgia, USA.
Groups:
- Rabies Vaccine With Antibiotics: Participants in this group received the rabies vaccines as well as an antibiotic regimen consisting of metronidazole, vancomycin, and neomycin sulfate.
- Rabies Vaccine: Participants in this group received the rabies vaccine.
Period: Overall Study
Arm/Group | Rabies Vaccine With Antibiotics | Rabies Vaccine
Started | 19 | 18
Completed (Completed the Day 28 assessment) | 14 | 15
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Early termination from study | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabies Vaccine With Antibiotics | Rabies Vaccine | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.42 (7.75) | 32.50 (6.58) | 32.46 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titers
Description: Antibody titers are examined by direct comparison of antibody titers in the blood. Rabies specific Immunoglobulin G (IgG) endpoint titer was measured by ELISA. The endpoint titer is defined as the reciprocal of the highest plasma dilution that gives a reading above the cutoff values. The cutoff is set based on the average plus 3 times the standard deviation of the reading of 1:160 dilution of baseline plasma.
Time Frame: Day 28
Population: This analysis includes participants who completed the Day 28 study visit.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Rabies Vaccine With Antibiotics | Rabies Vaccine
Number analyzed (Participants) | 14 | 15
IU/mL | 217.39 (262.99) | 805.64 (943.85)

2. Primary Outcome: Proportion of Participants Achieving Seroprotection
Description: Participants are categorized as achieving seropositivity if rabies specific IgG endpoint titer is present.
Time Frame: Day 28
Population: This analysis includes participants who completed the Day 28 study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Rabies Vaccine With Antibiotics | Rabies Vaccine
Number analyzed (Participants) | 14 | 15
Participants | 14 | 15

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time when the study intervention began through Day 56 of the study.
Arm/Group | Rabies Vaccine With Antibiotics | Rabies Vaccine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 2/19 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabies Vaccine With Antibiotics (N=19) | Rabies Vaccine (N=18)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03557008/Prot_SAP_000.pdf